CLINICAL TRIAL: NCT04692389
Title: The Efficacy of the Medical Device Jalosome® Soothing Gel in the Healing of Grade of 2 or 3 Radiodermatitis, Pain Intensity Reduction, as Well as Improvement of QoL in Oncology Patients: a Pilot Study.
Brief Title: Jalosome® Soothing Gel Efficacy Grade 2 or 3 Radiodermatitis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties in patients recruitment
Sponsor: Welcare Industries SpA (Industry)
Collaborators: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Welcare 012020
Record Dates: First submitted 2020-12-29; First posted 2020-12-31 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Radiodermatitis; Oncology; Quality of Life; Pain
Keywords: radiodermatitis; oncology; quality of life; pain; wound healing
MeSH Terms: conditions — Radiodermatitis; Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: The investigators would like to involve 30 oncology patients with 2 or 3 grade radiodermatitis (based on RTOG score).
  All oncology diagnosis will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Jalosome® Soothing gel (Experimental): The medical device will be applied by the patient himself, after appropriate training carried out by the nurse, twice a day, in the quantity necessary to cover the lesion (0.2g of gel /16 cm2 of skin (one spray), repeated as many times as necessary to cover the entire lesion). The treatment will last 8 weeks.
  The medical device will be delivered in the quantity strictly necessary to carry out the therapies between visits, in order to monitor its use. Patients will be seen weekly by the nurse, in order to ensure the best continuity of care and promote adherence to the study. Patients will be asked to keep a weekly diary, in which they will report their level of pain, analgesic therapy and medication. Nurses will be available for telephone counselling, if necessary.
  Interventions: Device: Jalosome soothing gel

INTERVENTIONS:
Device: Jalosome soothing gel — This study has not got other intervention
  Other Names: No other intervention

SUMMARY:
Testing the efficacy of the Jalosome® Soothing gel in 2 or 3 grade radiodermatitis healing in oncological patients.

The investigators would like to know also the efficacy of the device on quality of life and pain.

DETAILED DESCRIPTION:
The overall objective of the study is to evaluate the efficacy of the class IIA medical device Jalosome® soothing gel in the healing of grade 2 or 3 radiodermatitis, in oncology patients undergoing radiotherapy treatment, during a 8-week observation period.

The secondary endpoints are radiodermatitis pain control and quality of life.

The investigators would like to involve 30 oncology patients. All oncology diagnosis will be included in this pilot study. The study will adopt a quasi-experimental design with one arm. The results will be used to determine the sample size for a clinical trial in which the class IIA medical device Jalosome® soothing gel will be compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with cancer* undergoing radiotherapy treatment
* Patients with grade 2 or 3 radiotherapy lesions who are naive to radiodermatitis treatment or unresponsive to previous treatment
* Patients who have given written informed consent
* Patients expected to be followed at the centre for at least 8 weeks
* Patients with Karnofsky Performance Status(KPS) scale ≥ 40

Exclusion Criteria:

* Patients with grade 1 and grade IV radiodermatitis
* Patients with known intolerance to the components in Jalosome® soothing gel
* Patients who have already received radiotherapy in the past on the irradiated area
* Patients with cognitive impairment that does not allow adequate compliance with the protocol
* Patients with brain metastases
* Pregnant or lactating patients
* Patients with KPS < 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or 3 radiodermatitis healing | 8 weeks
  The primary endpoint is the number of grade 2 or 3 radiodermatitis healed by the application of Jalosome® soothing gel during the observation period, out of the total number of patients treated. This endpoint will be assessed by photographic documentation of lesion improvement and healing and with the aid of the RGOT scale (which should regress from grade 2 or 3 to grade 0 or 1).
  The time to regression of the lesion will also be monitored on this same endpoint in order to establish the rate of efficacy of the product against grade 2 and 3 lesions.

SECONDARY OUTCOMES:
Pain quality and intensity | 8 weeks
  The first secondary endpoint will be the intensity and quality of pain, measured respectively by the NRS scale and by questions on the type of pain perceived (twinge, burning, pins, allodynia (i.e. a painful impulse following a harmless stimulus), cramp-like, piercing (stab-like)).
Skindex questionnaire - 16 for quality of life | at the beginning, after 4 weeks and after 8 weeks
  Quality of life will then be assessed as a second enpoint, using the Skindex questionnaire - 16

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute Of Southern Switzerland -radio oncology unit, Bellinzona, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No